CLINICAL TRIAL: NCT03911648
Title: The Efficacy of Bupivacaine Alone and in Combination With Lidocaine at Performing Caudal Block on Analgesia in Pediatric Patients Underwent Circumcision: A Historical Cohort Study
Brief Title: Analgesic Efficacy of Lidocaine Plus Bupivacaine Versus Bupivacaine Alone Caudally
Status: Completed | Type: Observational
Sponsor: Ayancık State Hospital (Other Government)
Responsible Party: Principal Investigator, Ayse Gulsah Atasever, Resident Anesthesiologist, Ayancık State Hospital
Other Study IDs: 2019/366
Record Dates: First submitted 2019-04-09; First posted 2019-04-11 (Actual); Last update posted 2019-04-11 (Actual); Status verified 2019-04

CONDITIONS: Anesthesia, Local
Keywords: Bupivacaine; Lidocaine; Caudal block; Pediatric urologic surgery
MeSH Terms: interventions — Bupivacaine; Lidocaine

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group B;: Patients had 0.5 ml.kg-1 bupivacaine 0.25% caudally, the maximum given volume was 20 ml. N=42
  Interventions: Drug: 0.5 ml.kg-1 bupivacaine 0.25%
- Group L;: Patients had 0.5 ml.kg-1 bupivacaine 0.25% with the addition of 3 mg/kg lidocaine 1% caudally, the maximum given volume was 20 ml. N=44
  Interventions: Drug: 0.5 ml.kg-1 bupivacaine 0.25% with the addition of 3 mg/kg lidocaine 1%

INTERVENTIONS:
Drug: 0.5 ml.kg-1 bupivacaine 0.25% — Caudally
  Other Names: Marcaine
  Groups: Group B;
Drug: 0.5 ml.kg-1 bupivacaine 0.25% with the addition of 3 mg/kg lidocaine 1% — Caudally
  Other Names: Marcaine, Xylocaine
  Groups: Group L;

SUMMARY:
Optimal analgesia following ambulatory surgery is an important matter for patient satisfaction and it reduces unnecessary hospital admissions. This study investigated whether caudal block with different combinations of local anesthetics can alter postoperative pain scores and additional rescue analgesic use. The investigators also aim to determine the side effects of these technique such as nausea, vomiting, bradycardia, hypotension, respiratory depression, length of hospital stay, first micturition or mobilization times, surgical and anesthetic complications.

DETAILED DESCRIPTION:
Circumcision, which is performed on an outpatient basis is commonly a short durational operation in boys. Postoperative pain and agitation are the most common complaints in children with circumcision. The most important factor affecting the length of hospital stay is to provide an effective analgesia. Various methods are being used to manage postoperative pain such as caudal block, penile block, topical analgesia or intra-venous (iv) analgesics. Caudal block is applicable widely in pediatric day case surgery, providing excellent postoperative analgesia and attenuation of the stress response in children. Opioids can cause several side effects such as respiratory depression, suppression of bowel movements, nausea, vomiting, itching, addiction. Opioid drugs are not recommended in children as well. Lower abdominal surgeries affect dermatomes T10-L1 and blocking these nerve roots provides effective postoperative analgesia. Neuraxial blocks such as epidural and caudal blocks is considered the gold standard regional technique for pain management after lower abdominal surgery, blocking both somatic and visceral pain. Recent studies suggest that lidocaine and bupivacaine can be used in combination or a sole agent when performing regional anesthesia in children. But it remains unknown whether these combinations are useful or simply reflect underlying status. There is no report comparing the effects of bupivacaine alone and in combination with lidocaine at performing caudal epidural block in children. The investigators thus tested the primary hypothesis that combining the two different local anesthetics has a synergistic analgesic effect and can accelerate the onset time and decrease the need for additional analgesic doses. Secondarily, the investigators tested the hypothesis that providing intra-operative and postoperative analgesia reduces the risk of hemodynamic deteriorations, length of hospital stay, first micturition and mobilization times, surgical and anesthetic complications.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiologists (ASA) class 1.
* Patient underwent elective circumcision operation under general anesthesia and caudal analgesia.

Exclusion Criteria:

* Procedures simultaneously underwent another operation unrelated to circumcision.
* Patients who had unsuccessful caudal block.

Ages: 2 Years to 11 Years | Sex: Male
Age Groups: Child
Study Population: The medical records of pediatric patients who underwent circumcision under general anethesia with caudal block over 6 months (01 January 2018-31 June 2018) were analysed.
Sampling Method: Probability Sample
Enrollment: 86 (Actual)
Dates: Start 2018-07-01 (Actual); Primary Completion 2018-07-15 (Actual); Study Completion 2018-08-15 (Actual)

PRIMARY OUTCOMES:
Number of patients who require rescue analgesic | up to 10 hours
  iv/po analgesic use
The average pain scores | up to 10 hours
  Pain scores were typically recorded on a scale from 0 to 10 by visual analogue scale (VAS), whereas, in children younger than 4 years the FLACC (Face, Legs, Activity, Cry, Consolability) score was used.

SECONDARY OUTCOMES:
Number of participants with hypotension or bradycardia. | up to 10 hours
  An intra-operative decrease in blood pressure(BP) or heart rate(HR) of more than 20% from preoperative values was defined as hypotension or bradycardia, respectively, and was treated with rapid infusion of fluids or with atropine 0.01 mg/kg.
Number of participants with hypertension or tachycardia. | up to 10 hours
  An intraoperative increase in BP or HR by more than 20% was defined as insufficient analgesia and was treated with fentanyl 1 mcg/kg iv.
Incidence of side effects | up to 10 hours
  Nausea, vomiting, respiratory depression
Time to first mobilization | up to 10 hours
  Time to first mobilization
Time to first micturition | up to 10 hours
  Time to first micturition
The length of hospital stay | up to 10 hours
  Hospitalisation, hr

CONTACTS AND LOCATIONS:
Overall Officials: ayse gulsah atasever, MD, Principal Investigator — Ayancık State Hospital
Locations (1):
- Ayancık State Hospital, Sinop, Turkey (Türkiye)

REFERENCES:
- [Derived] Atasever AG, Ermis O, Demir BS, Kasali K, Karadeniz MS. Comparison of bupivacaine alone and in a combination with lidocaine for caudal block in patients undergoing circumcision: A historical cohort study. Turk J Urol. 2019 Nov 29;46(3):243-248. doi: 10.5152/tud.2019.19191. Print 2020 May. PMID 32401707
- See also: Brennan J. Modern day-case anaesthesia for children. Br J Anaesth. 1999;83:91-103. — https://www.ncbi.nlm.nih.gov/pubmed/?term=1.%09Brennan+LJ.+Modern+day-case+anaesthesia+for+children.+Br+J+Anaesth.+1999%3B83%3A91-103.
- See also: Suresh S et al. Are Caudal Blocks for Pain Control Safe in Children? An Analysis of 18,650 Caudal Blocks from the Pediatric Regional Anesthesia Network (PRAN) Database. Anesth Analgesia. 2015;120:151-156 — https://www.ncbi.nlm.nih.gov/pubmed/?term=Are+Caudal+Blocks+for+Pain+Control+Safe+in+Children%3F+An+Analysis+of+18%2C650+Caudal+Blocks+from+the+Pediatric+Regional+Anesthesia+Network+(PRAN)+Database.+Anesth+Analg.+2015%3B
- See also: Nancy B et al. Regional anesth and Pain Management for the Pediatric Patient. ınternatıonal anesthesıology clınıcs:2012; 50,4,83-95 — https://www.semanticscholar.org/paper/Regional-anesthesia-and-pain-management-for-the-Samol-Furstein/63c57069b2fe3354f6c78d4d7d08c8a550b7868a
- See also: Corliss A, Alyssa A, Timothy J, Danielle A Hamilton. Buffered lidocaine and bupivacaine mixture - the ideal local anesthetic solution? Plast Surg 2015: 23; 2, 87-90 — https://www.ncbi.nlm.nih.gov/pmc/articles/PMC4459414/